CLINICAL TRIAL: NCT01378143
Title: A Phase II Clinical Study Using OCZ103-OS in Patients With Unresectable and Locally Recurrent or Metastatic Colorectal Cancer Undergoing Standard Chemotherapy (mFOLFOX6 or FOLFIRI) as Second-Line Treatment
Brief Title: Using OCZ103-OS in Patients With Unresectable and Locally Recurrent or Metastatic Colorectal Cancer Undergoing Standard Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncozyme Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OP-103-C
Record Dates: First submitted 2011-06-15; First posted 2011-06-22 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2013-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Pentamidine bis(2-hydroxyethanesulfonate); OCZ103-OS; Standard of Care
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OCZ103-OS, mFOLFOX6 or FOLFIRI (Experimental): OCZ103-OS in combination with mFOLFOX6 or FOLFIRI as standard of care
  Interventions: Drug: OCZ103-OS [pentamidine bis(2-hydroxyethanesulfonate)], mFOLFOX6 or FOLFIRI

INTERVENTIONS:
Drug: OCZ103-OS [pentamidine bis(2-hydroxyethanesulfonate)], mFOLFOX6 or FOLFIRI — OCZ103-OS is given in combination with Chemotherapy each cycle

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of the use of OCZ103-OS in combination with standard of care as a second line treatment in subjects with unresectable and locally recurrent or metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a single arm, open label study to investigate the safety and efficacy of the use of OCZ103-OS in combination with standard therapy (mFOLFOX6 or FOLFIRI) as a second line treatment in subjects with unresectable and locally recurrent or metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven diagnosis of adenocarcinoma of the colon/rectum with evidence of (1) unresectable and, locally recurrent, or (2) metastatic disease.
2. Failure of first-line therapy(5-Fu-based therapy +/- bevacizumab) for metastatic colorectal cancer.
3. At least one (1) unidimensionally measurable lesion (on spiral CT scan).
4. 18 years of age or older.
5. ECOG performance status 0, 1 or 2.
6. Serum aspartate transaminase (AST), serum alanine transaminase (ALT), serum alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN), or AST,ALT, ALP ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
7. Total serum bilirubin ≤ 1.5 x ULN
8. Lipase and amylase within normal limits or abnormal limits but deemed not clinically significant.
9. Absolute neutrophil count (ANC) ≥ 1500/µL (1.5 x 10e9/L)
10. Platelets ≥ 100,000/µL (100 x 10e9/L)
11. Hemoglobin ≥ 90 g/L
12. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 60 ml/min. The Cockcroft-Gault formula to be used is as follows:

    eCcr=(140-age)x Mass(in kilogram)x Constant/Serum Creatinine(in µmol/L)

    Where Constant is 1.23 for men and 1.04 for women.
13. Normal or abnormal ECG. If ECG shows abnormalities, they must be deemed not clinically significant.
14. Signed and dated Informed Consent Form indicating that the subject (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
15. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures.
16. Life expectancy, in the opinion of the investigator, > 3 months.

Exclusion criteria

1. Systolic Blood Pressure <100 mmHg (if deemed clinically significant by the treating physician).
2. Uncontrolled diabetes, severe renal impairment or pancreatitis.
3. Concomitant therapy with other investigational agents or participation in another clinical trial within 30 days prior to enrollment.
4. Any of the following conditions: Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2; atrial fibrillation of any grade; QTc interval > 450 msec for males or > 470 msec for females or uncontrolled intercurrent illness, e.g. unstable angina; severe coronary disease, ventricular arrhythmias, bradycardia < 50 bpm; a history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia or family history of Long QT Syndrome).
5. Active uncontrolled bacterial infection.
6. Concurrent use of drugs that could prolong QT interval (NB: pentamidine is known to induce torsades de pointes) (see Appendix II: List of drugs that could prolong QT interval / we also suggest that you refer to the following link: http://www.azcert.org/medical-pros/drug-lists/bycategory.cfm).
7. Concurrent use of nephrotoxic drugs (depending on the medical health status of the patient and based on the judgment of the investigator), including but not limited to aminoglycosides, ampho B, foscarnet and cidofovir.
8. Concurrent use of drugs such as Rifampine and Lamivudine, since these that may be associated with pancreatitis.
9. Prior malignancy other than colorectal cancer (except for adequately treated carcinoma in situ of the cervix, non-melanoma skin cancer or localized prostate cancer with undetectable PSA level) unless the prior malignancy was diagnosed and definitively treated at least five (5) years previously with no subsequent evidence of recurrence.
10. Clinically significant non-malignant lung disease.
11. History of allergy or hypersensitivity to pentamidine.
12. Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to first dose of study medication.
13. Severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgement of the investigator, excess risk associated with trial participation of study drug administration, or which in the judgement of the investigator, would make the subject inappropriate for entry into this trial.
14. Use of oral anticoagulants (LMWH is acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Tumor size (CT scan) | 2 years
  To assess the antitumor activity of OCZ103-OS in combination with standard of care in subjects with unresectable and locally recurrent or metastatic colorectal cancer in terms of tumor growth during treatment
Progression free survival (PFS) | 2 years
  To assess the antitumor activity of OCZ103-OS in combination with standard of care in subjects with unresectable and locally recurrent or metastatic colorectal cancer in terms of progression free survival
Overall survival (OS) | 2 years
  To assess the antitumor activity of OCZ103-OS in combination with standard of care in subjects with unresectable and locally recurrent or metastatic colorectal cancer in terms of overall survival

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of OCZ103-OS | 2 months
  * To assess the peak plasma concentration of OCZ103-OS after administration on day 1 of first cycle.
  * Amount of OCZ103-OS in serum on day 1 of first cycle.
Number of participants with Adverse Events (AE) as a Measure of Safety and Tolerability | 2 years
  - To assess the number of adverse events in participants due to IV OCZ103-OS in conjunction with standard chemotherapy (mFOLFOX6- or FOLFIRI-contained regimen) in patients with unresectable and locally recurrent or metastatic colorectal cancer requiring second-line chemotherapy from baseline.
Objective response (OR) | 2 years
  - To assess the effect of OCZ103-OS on overall objective response (OR) in subjects with unresectable and locally recurrent or metastatic colorectal cancer treated concurrently with mFOLFOX6 or FOLFIRI.
Duration of response (DR) | 2 years
  - To assess the effect of OCZ103-OS on duration of response (DR) in subjects with unresectable and locally recurrent or metastatic colorectal cancer treated concurrently with mFOLFOX6 or FOLFIRI.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Kavan, MD, Ph.D., Principal Investigator — Jewish General Hospital; Benoit Samson, MD, Principal Investigator — CSSS Champlain - Charles-Lemoyne Hospital; Richard Letourneau, MD, Principal Investigator — St. Luc Hospital; Felix Couture, MD, Principal Investigator — Hotel-Dieu de Quebec; Felix Couture, MD, Principal Investigator — CSSS Alphonse-Desjardins; Annie Beaudoin, M.D., Principal Investigator — CHUS-Centre de recherche Etienne-Le Bel; Jacques Jolivet, MD, Principal Investigator — CSSS St-Jérome
Locations (7):
- Canada (7):
  - CSSS Champlain - Charles-Lemoyne Hospital, Greenfield Park, Quebec
  - CSSS Alphonse-Desjardins (CHAU Hotel-Dieu de Levis), Lévis, Quebec
  - CHUM-St. Luc Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
  - CHUS-Centre de recherche Etienne-Le Bel, Sherbrooke, Quebec
  - CSSS St-Jérome, St-Jérome, Quebec